CLINICAL TRIAL: NCT04761471
Title: Investigating the Role of Brain Oscillations in Reward-guided Behavior
Brief Title: Oscillations in Reward-guided Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Principal Investigator, Rafael Polania, Principal Investigator, Swiss Federal Institute of Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TI_Reward
Record Dates: First submitted 2021-02-05; First posted 2021-02-21 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Reward-guided Behaviour
Keywords: Brain oscillations; Neural oscillations; Transcranial electrical stimulation tCS; Temporal Interference stimulation TI; Decision-making

STUDY DESIGN:
Intervention Model Description: The same participants receive placebo/sham stimulation and active stimulation on different sessions separated with 1 week or within the same session.
  The sequence of sham/placebo and active stimulation will be randomized.
Masking Description: Participants will be not informed which stimulation they receive active or placebo/sham. They will be debriefed at the end of the experiment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TI stimulation (Experimental): Temporal interference (TI) stimulation is a type of low-intensity transcranial electrical stimulation with alternating current (tACS). In case of TI stimulation, 2 electric fields in kHz range are delivered to 4 electrodes, which are placed on the surface of the skull, to modulate neural oscillations.
  Interventions: Device: TI transcranial electrical stimulation

INTERVENTIONS:
Device: TI transcranial electrical stimulation — Participants will undergo transcranial electrical stimulation, which will be delivered with low current amplitudes (<= 2 mA) established with international safety guidelines for electrical stimulation. Threshold for the current amplitude will be established by participants themselves, such that they cannot distinguish when stimulation is applied and not applied.
  Duration of stimulation will not last longer than 30 minutes.

SUMMARY:
While people are reading, talking or playing computer games, their brain cells elicit electrical signals so they could perform these actions. The firing of these cells is not random but is organized in a temporal pattern, such that a group of cells are simultaneously active at a particular frequency. The researchers can read the frequency of brain signals and identify their location using different brain-imaging tools like EEG and fMRI. These methods are applied to healthy individuals and do not pose any danger.

The investigators of this project would like to use these techniques to study the brain signals, while healthy participants are making the decisions choosing between 2 rewards, e.g., 2 food items. Participants who have depression show different behavior while performing decision-making tasks and the investigation of processes that underlie them will lead to a better understanding of this disease.

Furthermore, there is another category of tools, which help to study the brain. This category includes electrical stimulation, which mimics the electrical pattern that brain cells elicit. Application of external electrical stimulation can enhance this pattern or disrupt it and this process will affect the behavior of a person. Recent investigations have led to the development of a new stimulation technique that allows targeting deep brain regions. The investigators of this project want to apply this method to change the performance of healthy participants in the tasks on decision-making. If this experiment is successful, then stimulation can be used as a therapy for participants with depression.

ELIGIBILITY:
General Inclusion Criteria:

* signed informed consent
* Age 18-40 years
* Normal physical and mental status (i.e. no neurological, musculoskeletal, neuromuscular, cognitive, or psychiatric disorders)
* If a participant already took part in the experiment with the same decision-making task

Exclusion Criteria for TI electrical stimulation:

* pregnancy
* epilepsy
* head traumas
* implants (cochlear, neurostimulators, cardiac pacemakers, medication infusion device)
* metal in the brain or skull
* work in the metal industry
* scars or inflammations on the regions, where the stimulation electrodes are placed
* administration of antipsychotic or anti-epileptic medication
* hearing problems or ringing in the ears
* syncope or fainting spells in the last 5 years
* severe side-effects after transcranial magnetic stimulation (TMS) or electrical stimulation if participant underwent it before
* the inability to comply with magnetic resonance imaging (MRI) inclusion criteria if participant underwent it before

Exclusion Criteria for MRI experiments:

* pregnancy
* claustrophobia
* history of brain surgery
* family member that suffers from epilepsy
* suffering from medication abuse for more than a year or drug intake
* taking medications for medical reasons for more than a month
* receiving of depot injections
* one or more of the following materials in the body: metallic objects (e.g., dental implants, a metallic splinter in the eye, but not braces); wire, pacemaker or implanted defibrillator; artificial heart valves; vascular grafts; bio-stimulator or nerve stimulator; aneurysm or intracranial clip; cochlear implant; other prostheses or orthoses; implanted medication pump (insulin or pain pump); medicated patch (e.g., nitro-patch, pain patch, nicotine patch, hormone patch, motion sickness patch); other implants; tattoo or jewelry
* history of any of these illnesses: brain thrombosis, stroke, traumatic brain injury, meningitis, heart attack, prolonged loss of consciousness, migraine, epilepsy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2023-12-04 (Actual)

PRIMARY OUTCOMES:
Accuracy | Continuously while participants perform a cognitive task (circa 2 hours) with and without TI stimulation.
  Accuracy will be collected with a keyboard and a mouse
Reaction time | Continuously while participants perform a cognitive task (circa 2 hours) with and without TI stimulation.
  Reaction time will be collected with a keyboard and a mouse
Fixations | Continuously while participants perform a cognitive task (circa 2 hours) with and without TI stimulation.
  Fixations of the gaze on the screen will be recorded with an eye-tracker.
Saccades | Continuously while participants perform a cognitive task (circa 2 hours) with and without TI stimulation.
  Saccades (a type of the eye movement) will be recorded with an eye-tracker.
Blood oxygenation level dependent (BOLD) | Continuously while participants perform a cognitive task (circa 2 hours) with and without TI stimulation.
  BOLD signal is measured with functional magnetic resonance imaging (fMRI) experiment.
Brain oscillations in delta band | Continuously while participants perform a cognitive task (circa 2 hours) with and without TI stimulation.
  Oscillations within the range from 0.5 Hz to 4 Hz will be measured with electroencephalography (EEG).
Brain oscillations in theta band | Continuously while participants perform a cognitive task (circa 2 hours) with and without TI stimulation.
  Oscillations within the range from 4 Hz to 8 Hz will be measured with EEG.
Brain oscillations in alpha band | Continuously while participants perform a cognitive task (circa 2 hours) with and without TI stimulation.
  Oscillations within the range from 8 Hz to 12 Hz will be measured with EEG.
Brain oscillations in beta band | Continuously while participants perform a cognitive task (circa 2 hours) with and without TI stimulation.
  Oscillations within the range from 12 Hz to 30 Hz will be measured with EEG.
Brain oscillations in low gamma band | Continuously while participants perform a cognitive task (circa 2 hours) with and without TI stimulation.
  Oscillations within the range from 30 Hz to 70 Hz will be measured with EEG.
Brain oscillations in high gamma band | Continuously while participants perform a cognitive task (circa 2 hours) with and without TI stimulation.
  Oscillations within the range from 70 Hz to 250 Hz will be measured with EEG.

OTHER OUTCOMES:
Safety outcome (Headache) | This outcome will be recorded after each experiment with TI stimulation. One experiment lasts around 2 hours. These experiments will be held with different participants throughout the whole study (around 3 years).
  Headache severity will be collected with a questionnaire that contains a scale on which participant can rate this side-effect: (1) absent, (2) mild, (3) moderate, (4) severe. After this question, participant is asked to estimate relationship of this side-effect to intervention: (1) none, (2) remote, (3) possible, (4) probable, (5) definite.
Safety outcome (Scalp pain) | This outcome will be recorded after each experiment with TI stimulation. One experiment lasts around 2 hours. These experiments will be held with different participants throughout the whole study (around 3 years).
  Scalp pain severity will be collected with a questionnaire that contains a scale on which participant can rate this side-effect: (1) absent, (2) mild, (3) moderate, (4) severe. After this question, participant is asked to estimate relationship of this side-effect to intervention: (1) none, (2) remote, (3) possible, (4) probable, (5) definite.
Safety outcome (Tingling) | This outcome will be recorded after each experiment with TI stimulation. One experiment lasts around 2 hours. These experiments will be held with different participants throughout the whole study (around 3 years).
  Tingling severity will be collected with a questionnaire that contains a scale on which participant can rate this side-effect: (1) absent, (2) mild, (3) moderate, (4) severe. After this question, participant is asked to estimate relationship of this side-effect to intervention: (1) none, (2) remote, (3) possible, (4) probable, (5) definite.
Safety outcome (Itching) | This outcome will be recorded after each experiment with TI stimulation. One experiment lasts around 2 hours. These experiments will be held with different participants throughout the whole study (around 3 years).
  Itching severity will be collected with a questionnaire that contains a scale on which participant can rate this side-effect: (1) absent, (2) mild, (3) moderate, (4) severe. After this question, participant is asked to estimate relationship of this side-effect to intervention: (1) none, (2) remote, (3) possible, (4) probable, (5) definite.
Safety outcome (Burning) | This outcome will be recorded after each experiment with TI stimulation. One experiment lasts around 2 hours. These experiments will be held with different participants throughout the whole study (around 3 years).
  Burning sensations will be collected with a questionnaire that contains a scale on which participant can rate this side-effect: (1) absent, (2) mild, (3) moderate, (4) severe. After this question, participant is asked to estimate relationship of this side-effect to intervention: (1) none, (2) remote, (3) possible, (4) probable, (5) definite.
Safety outcome (Discomfort) | This outcome will be recorded after each experiment with TI stimulation. One experiment lasts around 2 hours. These experiments will be held with different participants throughout the whole study (around 3 years).
  Discomfort sensations will be collected with a questionnaire that contains a scale on which participant can rate this side-effect: (1) absent, (2) mild, (3) moderate, (4) severe. After this question, participant is asked to estimate relationship of this side-effect to intervention: (1) none, (2) remote, (3) possible, (4) probable, (5) definite.
Safety outcome (Nausea) | This outcome will be recorded after each experiment with TI stimulation. One experiment lasts around 2 hours. These experiments will be held with different participants throughout the whole study (around 3 years).
  Nausea sensations will be collected with a questionnaire that contains a scale on which participant can rate this side-effect: (1) absent, (2) mild, (3) moderate, (4) severe. After this question, participant is asked to estimate relationship of this side-effect to intervention: (1) none, (2) remote, (3) possible, (4) probable, (5) definite.
Safety outcome (Fatigue) | This outcome will be recorded after each experiment with TI stimulation. One experiment lasts around 2 hours. These experiments will be held with different participants throughout the whole study (around 3 years).
  Fatigue sensations will be collected with a questionnaire that contains a scale on which participant can rate this side-effect: (1) absent, (2) mild, (3) moderate, (4) severe. After this question, participant is asked to estimate relationship of this side-effect to intervention: (1) none, (2) remote, (3) possible, (4) probable, (5) definite.
Safety outcome (Acute mood change) | This outcome will be recorded after each experiment with TI stimulation. One experiment lasts around 2 hours. These experiments will be held with different participants throughout the whole study (around 3 years).
  Acute mood change will be collected with a questionnaire that contains a scale on which participant can rate this side-effect: (1) absent, (2) mild, (3) moderate, (4) severe. After this question, participant is asked to estimate relationship of this side-effect to intervention: (1) none, (2) remote, (3) possible, (4) probable, (5) definite.
Safety outcome (Phosphenes) | This outcome will be recorded after each experiment with TI stimulation. One experiment lasts around 2 hours. These experiments will be held with different participants throughout the whole study (around 3 years).
  Phosphenes/light sensations will be collected with a questionnaire that contains a scale on which participant can rate this side-effect: (1) absent, (2) mild, (3) moderate, (4) severe. After this question, participant is asked to estimate relationship of this side-effect to intervention: (1) none, (2) remote, (3) possible, (4) probable, (5) definite.
Safety outcome (Sleeplessness) | This outcome will be recorded after each experiment with TI stimulation. One experiment lasts around 2 hours. These experiments will be held with different participants throughout the whole study (around 3 years).
  Sleeplessness will be collected with a questionnaire that contains a scale on which participant can rate this side-effect: (1) absent, (2) mild, (3) moderate, (4) severe. After this question, participant is asked to estimate relationship of this side-effect to intervention: (1) none, (2) remote, (3) possible, (4) probable, (5) definite.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Polania, PhD, Principal Investigator — ETH Zürich
Locations (1):
- ETH Zurich, Zurich, Schweiz, Switzerland

IPD SHARING:
Plan to Share IPD: No